CLINICAL TRIAL: NCT00352547
Title: Influence of MDR-1 CYP3A4 and CYP3A5 Genotypes/Haplotypes on Sirolimus Pharmacokinetics and Pharmacodynamics in Patients With Renal Transplantation
Brief Title: Influence of Genes on Sirolimus Metabolism in Patients With Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040184; 04-CC-0184
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-12-02

CONDITIONS: Renal Transplant
Keywords: Immunosuppresant; Genetic Polymorphism; Drug Metabolism; Pharmacogenetics; Rapamycin

SUMMARY:
This study will evaluate the effects of certain genes (MDR-1, CYP3A4, and CYP3A5) on metabolism of the drug sirolimus, an immune-suppressing drug given to transplant recipients to prevent organ rejection. Individual differences in metabolism and excretion of sirolimus affect the patient's response to treatment.

Patients who have undergone kidney transplantation at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Transplant Branch and have received sirolimus treatment will be enrolled in this study.

DNA (genetic material) will be extracted from blood samples collected from transplant recipients to determine their MDR-1, CYP3A4, and CYP3A5 genotypes. Patient demographic information and data on sirolimus metabolism and excretion will be collected from the medical information system, NIDDK transplant database, and the patients' medical records. The data will be compared among patients with different genotypes (genetic constitution of an individual) and haplotypes (set of genes that code for different proteins but are inherited as a unit) to determine the effect of these gene variations on sirolimus metabolism.

Information from this study may be applied to developing better dosing strategies, and thus, treatment outcomes for transplant patients receiving sirolimus.

DETAILED DESCRIPTION:
The immunosuppressant sirolimus is a substrate for the drug efflux pump p-glycoprotein

(Pgp) and the hepatic and intestinal drug metabolizing enzyme cytochrome P450 3A4/5

(CYP3A4/5). Single nucleotide polymorphisms (SNPs) in the multi-drug resistance (MDR)-1

gene which encodes for the Pgp, CYP3A4, and CYP3A5 genes have been shown to be associated with altered metabolism of various drugs including the immunosuppressants cyclosporine and tacrolimus. This protocol will evaluate the effects of MDR-1, CYP3A4, and CYP3A5 gentotypes/haplotypes on the pharmacokinetics and pharmacodynamics of sirolimus in patients with renal transplantation. All patients who had kidney transplantation at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Transplant Branch, participated in one of the NIDDK therapeutic protocols, and have received sirolimus will be enrolled in this study. Selected MDR-1, CYP3A4, and CYP3A5 SNPs will be determined by polymerase chain reaction based methods using existing patient blood samples. Demographic, pharmacokinetic, and pharmacodynamic data will be collected from the medical information system, NIDDK transplant database, and medical records of these patients. Population pharmacokinetic parameters and pharmacodynamic measurements will then be compared among patients with different MDR-1, CYP3A4, and CYP3A5 genotypes/haplotypes. Results from this study will help to understand the effects of pharmacogenetics on sirolimus pharmacokinetics and pharmacodynamics, and will provide information for rationalizing sirolimus dosing in patients with renal transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who meet the following criteria will be included in the study:

* Underwent kidney transplantation at the NIDDK Transplant Branch; and
* Participated in one of the NIDDK therapeutic protocols, and
* Have received or switched to sirolimus

EXCLUSION CRITERIA:

Patients with clearly documented non-compliance to medications including sirolimus will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-05-21; Study Completion 2013-12-02

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Penzak, Pharm.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sattler M, Guengerich FP, Yun CH, Christians U, Sewing KF. Cytochrome P-450 3A enzymes are responsible for biotransformation of FK506 and rapamycin in man and rat. Drug Metab Dispos. 1992 Sep-Oct;20(5):753-61. PMID 1385058
- [Background] Ferron GM, Mishina EV, Zimmerman JJ, Jusko WJ. Population pharmacokinetics of sirolimus in kidney transplant patients. Clin Pharmacol Ther. 1997 Apr;61(4):416-28. doi: 10.1016/S0009-9236(97)90192-2. PMID 9129559
- [Background] Kahan BD, Napoli KL, Kelly PA, Podbielski J, Hussein I, Urbauer DL, Katz SH, Van Buren CT. Therapeutic drug monitoring of sirolimus: correlations with efficacy and toxicity. Clin Transplant. 2000 Apr;14(2):97-109. doi: 10.1034/j.1399-0012.2000.140201.x. PMID 10770413